CLINICAL TRIAL: NCT00953030
Title: Cost Effective Health Promotion for Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Susan L. Hughes, Center for Research on Health and Aging, University of Illinois Chicago
Allocation: Randomized | Masking: None
Other Study IDs: R01DP000094 (NIH)
Record Dates: First submitted 2009-08-05; First posted 2009-08-06 (Estimated); Last update posted 2009-08-06 (Estimated); Status verified 2009-08

CONDITIONS: Working Adults

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- COACH (Experimental): web-based risk assessments with an action plan that is negotiated with a "Coach" who provides personalized follow-up reinforcement
  Interventions: Behavioral: COACH
- RealAge (Experimental): a web-based health risk assessment and risk profile with disease-specific follow-up reinforcement modules
  Interventions: Behavioral: RealAge
- light health education control (No Intervention)

INTERVENTIONS:
Behavioral: COACH
  Arms: COACH
Behavioral: RealAge
  Arms: RealAge

SUMMARY:
This project tests the cost-effectiveness of two promising evidence-based health promotion/ behavior change interventions. The first intervention is the COACH Program, a revised version of the Health Enhancement Program (HEP) that has been implemented to date with older adults at multiple Senior Centers across the country (Leveille et al, 1998). The second is the web-based RealAge program which is also being implemented for older adults at multiple sites nationally and internationally. The Coach program combines a web-based risk assessment with individualized counselling. In contrast, RealAge is a totally web-based program.

The specific hypotheses that we will test in the proposed cost-effectiveness study are shown below.

Primary Study Hypotheses:

COACH participants will experience significantly greater reductions in absenteeism, disability days, and healthcare use and cost at 6 and 12 months than RealAge participants. Participants in both the COACH and RealAge treatment groups will experience significantly greater reductions in absenteeism, disability days, and healthcare use and cost than control group participants at 6 and 12 months.

Secondary Study Hypotheses:

COACH participants will experience significantly greater levels of adherence to health promotion Action Plans and greater reduction in weight, body mass index, blood pressure and depression and greater increase in vitality and quality of life than RealAge participants at 6 and 12 months. Participants in both the COACH and RealAge treatment arms will experience significantly better outcomes on these measures at 6 and 12 months than control group participants.

ELIGIBILITY:
Inclusion Criteria:

* Current employee of the University of Illinois at Chicago
* 40+ years of age

Exclusion Criteria:

* Those not currently employed by the University of Illinois at Chicago
* Those under the age of 40

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 423 (Actual)
Dates: Start 2004-09; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois Chicago, Chicago, Illinois, United States